CLINICAL TRIAL: NCT07068672
Title: Effect of Kaleidoscope and Helicone Use on Pain and Anxiety During Venipuncture in School-Age Children: A Randomized Controlled Trial
Brief Title: Kaleidoscope and Helicone for Pain and Anxiety in Children
Acronym: KHALPAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AYLİN ARIKAN (Other)
Responsible Party: Sponsor-Investigator, AYLİN ARIKAN, Doctor of Philosophy in Pediatric Nursing, Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AESH-B-2025-0123; AEŞH-BADEK-2025-0123 (Other: Ankara University)
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Pain Management; Procedural Pain; Children; Pediatric Nursing
Keywords: Kaleidoscope; Helicone; Pediatric Pain Management; School-Age Children; Venipuncture
MeSH Terms: conditions — Agnosia; Pain, Procedural

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kaleidoscope Group (Experimental): Children in this group were provided with a handheld kaleidoscope starting 2 minutes before and during venipuncture. The visual distraction created by the kaleidoscope's changing colorful patterns aimed to reduce pain and anxiety. The child focused on the visual display throughout the procedure.
  Interventions: Behavioral: Kaleidoscope
- Helicone Group (Experimental): Children in this group used a helicone toy starting 2 minutes before and during venipuncture. The toy, which changes shape with hand manipulation, provided active distraction to reduce pain and anxiety by engaging both visual and tactile senses.
  Interventions: Behavioral: Helicone
- Control Group (No Intervention): Children in this group received standard care during venipuncture without any distraction tools. No visual or tactile distraction was provided.

INTERVENTIONS:
Behavioral: Kaleidoscope — A handheld kaleidoscope was used as a passive distraction tool during venipuncture. The device was introduced to the child 2 minutes before the procedure and remained in view during blood collection. It provided dynamic, colorful visual stimuli to help reduce pain and anxiety.
  Arms: Kaleidoscope Group
Behavioral: Helicone — A helicone toy was used as an active distraction tool. Children held and rotated the device beginning 2 minutes before and during venipuncture. The interactive movement and shape-shifting design engaged the child's attention to reduce procedural pain and anxiety.
  Arms: Helicone Group

SUMMARY:
This randomized controlled trial aimed to evaluate the effects of kaleidoscope and helicone distraction tools on pain and anxiety levels during venipuncture in school-age children. The study was conducted at Ankara Etlik City Hospital Pediatric Emergency Department between April and May 2025. A total of 210 children aged 6 to 12 years who were undergoing venous blood sampling for the first time were randomly assigned to one of three groups: Kaleidoscope, Helicone, or Control (standard care). The Kaleidoscope group used a passive distraction tool featuring dynamic visual patterns; the Helicone group used an active distraction tool that involves hand manipulation of a rotating toy. Pain levels were measured using the Wong-Baker FACES Pain Rating Scale, and anxiety levels were assessed using the Children's Anxiety Meter-State (CAM-S). Measurements were taken before, during, and after the procedure. This study seeks to determine the comparative effectiveness of active versus passive distraction techniques in pediatric procedural pain and anxiety management. All interventions were non-pharmacological, non-invasive, and conducted in a safe clinical setting with informed consent obtained from both children and their guardians.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 6 and 12 years
* Requiring venipuncture for clinical purposes
* Able to verbally communicate pain and anxiety
* Accompanied by a parent or legal guardian who provides written informed consent
* Child provides verbal assent to participate

Exclusion Criteria:

* Children with cognitive or neurological disorders affecting pain or anxiety perception
* Use of any analgesics, anxiolytics, or sedatives within 6 hours prior to the procedure
* Visual or hearing impairments that interfere with the use of kaleidoscope or helicone
* Previous experience with similar distraction tools
* Presence of any skin condition preventing pain scale assessment

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Pain level measured using Wong-Baker FACES Pain Scale | Two minutes before the procedure, during needle insertion, and two minutes after the procedure
  Pain was assessed by the child using the Wong-Baker FACES Pain Rating Scale. This scale ranges from 0 to 10, where higher scores indicate more severe pain. Evaluations were conducted at three time points: before the procedure, during needle insertion, and two minutes after.
Anxiety level measured using Children's Anxiety Meter - State (CAM-S) | Two minutes before the procedure, during needle insertion, and two minutes after the procedure
  Anxiety was evaluated using the Children's Anxiety Meter - State (CAM-S) tool. The scale ranges from 0 (no anxiety) to 10 (extreme anxiety). Assessments were completed by the child with assistance from the researcher at three time points: before, during, and after the venipuncture.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No